CLINICAL TRIAL: NCT03267524
Title: Walking for Recovery From Surgery: Pilot Study of a Prehabilitation Intervention for Older Adults With Cancer and Their Family Caregivers
Brief Title: Walking for Recovery From Surgery in Improving Quality of Life in Older Adults With Lung or Gastrointestinal Cancer and Their Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17277; NCI-2017-01565 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Adult Liver Carcinoma; Caregiver; Colorectal Carcinoma; Lung Carcinoma; Malignant Digestive System Neoplasm; Pancreatic Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms; Lung Neoplasms; Gastrointestinal Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Walking for Recovery from Surgery) (Experimental): Patients and caregivers receive Walking for Recovery from Surgery prehabilitation intervention in 4 sessions 3-7 days before surgery, before discharge, and at 2 and 7 days post-discharge.
  Interventions: Behavioral: Exercise Intervention; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Receive Walking for Recovery from Surgery prehabilitation intervention
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Survey Administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies how well Walking for Recovery from Surgery works in improving quality of life in older adults with lung or gastrointestinal cancer and their family caregivers. A walking program, such as Walking for Recovery from Surgery may help support overall well-being as a caregiver, and may help improve family member or friend's recovery from surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine whether the intervention and telehealth approach would be feasible and acceptable.

SECONDARY OBJECTIVES:

I. To examine patient outcome patterns suggesting the potential efficacy of the intervention on self-efficacy, functional status (daily steps, 6-minute walk time, timed up and go), psychological distress, symptoms, and global health status.

OUTLINE:

Patients and caregivers receive Walking for Recovery from Surgery prehabilitation intervention in 4 sessions 3-7 days before surgery, before discharge, and at 2 and 7 days post-discharge.

After completion of study, patients and caregivers are followed up for 2 months.

ELIGIBILITY:
-Inclusion:

* PATIENT: Diagnosis of lung or GI (colorectal, pancreas, liver) cancers
* PATIENT: Scheduled to undergo surgery
* PATIENT: >= 65 years
* PATIENT: Able to read and understand English
* CAREGIVER: Family member/friend identified by the patient as the primary caregiver before and after surgery
* CAREGIVER: >= 21 years
* CAREGIVER: Able to read and understand English
* This study will be conducted in patients and family caregivers who are scheduled to undergo lung or GI cancer surgery treatment
* There are no restrictions related to performance status or life expectancy
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion

• Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Pedometer-assessed daily steps (patients) | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
6-minute walking time (patients) | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
Timed-up and go (patients) | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
Short Physical Performance Battery (patients) | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
General health status assessed using Patient-Reported Outcomes Measurement Information System (PROMIS) General Physical and Mental Health-Short Form (patients) | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
Symptoms (patients) | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
Distress level assessed using Distress Thermometer (patients) | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
Self-efficacy (caregivers) | Up to 2 months
  Will be assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy-Short Form. Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
Distress assessed using Distress thermometer (caregivers) | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
General health status assessed using Patient-Reported Outcomes Measurement Information System (PROMIS) General Physical and Mental Health-Short Form (caregivers) | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
Functional status (caregivers) | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.
Geriatric assessment | Up to 2 months
  Descriptive statistics will be used to summarize all outcome measure scores using validated scoring procedures, and to evaluate patterns suggesting potential intervention efficacy on outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, RN, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Lafaro KJ, Raz DJ, Kim JY, Hite S, Ruel N, Varatkar G, Erhunmwunsee L, Melstrom L, Lee B, Singh G, Fong Y, Sun V. Pilot study of a telehealth perioperative physical activity intervention for older adults with cancer and their caregivers. Support Care Cancer. 2020 Aug;28(8):3867-3876. doi: 10.1007/s00520-019-05230-0. Epub 2019 Dec 16. PMID 31845007